CLINICAL TRIAL: NCT01776814
Title: Comparison of the Efficacy of Entecavir and Tenofovir Monotherapy for the Treatment of Nucleos(t)Ide-naïve Patients With Chronic Hepatitis B in Korea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Ju Seung Kim, MD, principle investigator, Gachon University Gil Medical Center
Other Study IDs: GAIRB2963-2012
Record Dates: First submitted 2013-01-18; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Hepatitis B
Keywords: Entecair; Tenofovir
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic hepatitis B virus infection is an important cause of morbidity and mortality. Tenofovir disoproxil fumarate and entecavir were licensed for the treatment of hepatitis B virus infection. In this study, the investigators will try to make comparison between Entecavir and Tenofovir and investigate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 < Age < 70
* HBV DNA > 100,000 copies/mL and increased ALT over 2 times compared with normal range if HBsAg (+), HBeAg (+)
* HBV DNA > 10,000 copies/mL and increased ALT compared with normal range if HBsAg (+), HBeAg (-)

Exclusion Criteria:

* With HCV or other liver disease
* With kidney disease
* decompensated liver cirrhosis
* with hepatocellular carcinoma
* refuse this clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: treatment of nucleos(t)ide-naive patients who were diagnosed with chronic hepatitis B in Korea
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
virologic response | changes from baseline HBV DNA level at 3, 6, 9, 12 months after taking entecavir or tenofovir
  Patients will check the HBV DNA level at 3, 6, 9, 12 months after taking entecavir and tenofovir

SECONDARY OUTCOMES:
reduction of alanine transaminase | changes from baseline ALT level at 3,6,9,12 months after taking entecavir or tenofovir
  Patients will check the level of alanine transaminasel at 3, 6, 9, 12 months after taking entecavir and tenofovir

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Department of Gastroenterology, Incheon, South Korea